CLINICAL TRIAL: NCT01905176
Title: The Effectiveness of Multiple Nursing Interventions, for Promoting Heart Failure Self-care, on Patients' Quality of Life and Heart Failure Outcomes: A Randomized Control Trial.
Brief Title: Management of Patients With HF by Using Educational or Educational & Telephone or Telephone Interventions and Support in Cyprus
Acronym: MEETTinCY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyprus University of Technology (Other)
Collaborators: University of Athens (Other)
Responsible Party: Principal Investigator, Ekaterini Lambrinou, Assistant Professor, Cyprus University of Technology
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: MEETTinCY
Record Dates: First submitted 2013-07-15; First posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Randomized Control Trial; Disease management; Self-care; Nursing; Patient education as topic
MeSH Terms: conditions — Heart Failure | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Predischarge educational intervention (Experimental): In person education on heart failure topics before discharge
  Interventions: Other: In person education on heart failure topics before discharge
- Telephone educational intervention (Experimental): Telephone support and education post-discharge
  Interventions: Other: Telephone support and education post-discharge
- Combination (Experimental): Pre-discharge in person education and post-discharge telephone education and support
  Interventions: Other: Pre-discharge in person education and post-discharge telephone education and support
- Usual care (control group) (No Intervention): Patients receive the routine care provided by the hospital which does not involve protocol driven discharge-planning

INTERVENTIONS:
Other: In person education on heart failure topics before discharge — Individualized in-person education on HF topics aiming to promote self-care practices by using educational electronic material and booklet
  Arms: Predischarge educational intervention
Other: Telephone support and education post-discharge — Individualized telephone support/education of three months duration, on HF topics, aiming to promote self-care practices while evaluating patients' current status and condition
  Arms: Telephone educational intervention
Other: Pre-discharge in person education and post-discharge telephone education and support — Patients receive both interventions of Arm 1 & 2: individualized pre-discharge counseling/education along with telephone follow-up support for three months, following the same line as mentioned in Arms 1 & 2
  Arms: Combination

SUMMARY:
The current trial aims to examine the effectiveness of three different types of nursing interventions, on heart failure (HF) patients' quality of life and on HF outcomes, compared to the usual care. The interventions include promotion of self-care practices through education and support; they are either provided before discharge, post-discharge through telephone, or both.

DETAILED DESCRIPTION:
The current trial aims to examine the effectiveness of three different types of nursing interventions, on heart failure (HF) patients' quality of life and on HF outcomes, compared to the usual care. The interventions include promotion of self-care practices through education and support. HF patients admitted in the public hospitals of the Cyprus Republic are screened for eligibility. Consented patients who meet the inclusion criteria are recruited before their discharge, and are randomly allocated to one of the four groups of the trial. Patients of the three intervention groups receive educational intervention and support, before discharge or post-discharge through telephone, or both. Patients of the fourth group receive the usual care (control group). The patients' follow up period is 3 months. The main purpose of the study is to determine whether the combination of predischarge education/support and tele-management is more efficient in improving HF outcomes, rather than the in-person and telephonic components alone. Outcome measures include quality of life and HF events (re-admissions and death) and time to HF event.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patients with evidenced HF
* Planned for discharge
* NYHA class I-IV
* Greek speaking
* Able and willing to give informed consent

Exclusion Criteria:

* Severe mental illness or severly impaired cognitive function
* Patients that are to be transferred to nursing or rehabilitation homes
* Patients unable to be contacted via telephone
* Patients with active cancer
* Patients on dialysis
* Patients scheduled for surgery
* Patients recently undergone surgery (up to 3 months)
* Patients with less than 3 months life expectancy (end-stage)
* Patients with chronic degenerative diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in heart failure related quality of life at 3 months | 3 months
  Measuring the difference in quality of life scores from baseline to 3 months, by using a disease specific instrument for estimating quality of life in heart failure patients

SECONDARY OUTCOMES:
Change from baseline in heart failure self-care behavior at 3 months | 3 months
  Measuring the difference from baseline to 3 months, in self-care behavior scores by using a heart failure specific instrument
Combined outcome of readmission or death at 3 months post discharge | 3 months
  Number of participants presented with at least one event in terms of rehospitalization and / or death, during the 3 months follow up period
Change in heart failure knowledge from baseline to 3 months | 3 months
  Measuring the difference, from baseline to 3 months, in heart failure knowledge scores by using a heart failure specific instrument
Change from baseline in general health status (functioning) at 3 months | 3 months
  Measuring the change, from baseline to 3 months, in general health status (functioning), by using a non-disease specific instrument

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterini Lambrinou, Study Director — Cyprus University of Technology
Locations (1):
- Cyprus University of Technology; Nursing Department, Limassol, Limassol District, Cyprus

REFERENCES:
- [Derived] Lambrinou E, Protopapas A, Paikousis L, Middleton N, Papathanassoglou EDE, Sourtzi P, Kaloyirou F. Effectiveness of a multicentre randomized controlled trial with three different nurse-led intervention management programmes for patients with heart failure: the main results of the MEETinCY study. Eur J Cardiovasc Nurs. 2025 Mar 3;24(2):290-300. doi: 10.1093/eurjcn/zvae169. PMID 39873659